CLINICAL TRIAL: NCT02496806
Title: Seaweed Derived Anti-inflammatory Agents and Antioxidants
Brief Title: The Absorption and Metabolism of Seaweed Polyphenols in Humans
Acronym: SWAFAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: University of Ulster (Other)
Responsible Party: Principal Investigator, DR GIULIA CORONA, Dr., University of Reading
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SWAFAX11/18
Record Dates: First submitted 2015-06-24; First posted 2015-07-14 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
Keywords: Polyphenols; Absorption; Metabolism; Phlorotannins; Seaweeds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): 400mg capsule containing seaweed extract (treatment) Intervention: Dietary Supplement: Treatment capsule containing seaweed extract (treatment)
  Interventions: Dietary Supplement: Seaweed extract

INTERVENTIONS:
Dietary Supplement: Seaweed extract — Treatment capsule containing seaweed extract (treatment)

SUMMARY:
Brown seaweeds are a rich source of phlorotannins, a characteristic class of polyphenols which are unique to seaweeds of this type and can comprise 5 to 15 % of the dried weight. Unlike other classes of polyphenols, there is a lack of knowledge regarding phlorotannins and their bioavailability and bioactivity. The purpose of this study is to investigate the absorption and metabolism of seaweed polyphenols in humans. As part of an EC project (SWAFAX), an acute clinical intervention will be conducted to investigate the metabolism/ bioavailability of brown seaweed phlorotannins. Urine and plasma samples from 24 healthy volunteers that consumed a seaweed capsule containing polyphenols will be collected before and after the intervention. Data emanating from this project will provide strong scientific evidence for bioavailability and health promoting activity of a seaweed polyphenol extract in human volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Body Mass Index of 18-30 Kg/m2

Exclusion Criteria:

* Inability to swallow capsules
* Smoking
* Alcohol intake of >21 units/wk
* Blood pressure > 150/90 mmHg
* Any dietary restrictions or weight reducing diet
* Vegetarian
* Heamoglobin levels< 125 g/l for male, < 110 g/l for female,
* Gamma GT levels > 80 IU/l
* Cholesterol levels > 6.5 mmol/l
* Myocardial infarction or stroke in the previous 12 months
* Gastrointestinal disease or chronic gastrointestinal disorders
* Reproductive disorder
* Blood-clotting disorder
* Metabolic disorders
* Lipid-modifying medication
* Blood clotting mdication
* Antibiotic medication in previous 3 months before study
* Lactation
* Pregnancy
* Females of childbearing potential and not using effective contraceptive precautions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Seaweed polyphenol metabolites in urine | 24 hours
Seaweed polyphenol metabolites in plasma | 24 hours

SECONDARY OUTCOMES:
Citokine levels in plasma | 24 hours